CLINICAL TRIAL: NCT02544152
Title: A Randomized, Double-blind, Placebo-Controlled, Multicenter Study of the Efficacy and Safety of Lubiprostone in Adult Subjects With Mixed or Unsubtyped Irritable Bowel Syndrome (IBS-M/IBS-U)
Brief Title: Evaluation of the Efficacy and Safety of Lubiprostone in Adults With Mixed or Unsubtyped Irritable Bowel Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Sucampo Pharma Americas, LLC (Industry)
Collaborators: Takeda (Industry); Sucampo AG (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCMP-0211-201
Record Dates: First submitted 2015-08-20; First posted 2015-09-09 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2018-03

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Care provider and outcomes assessor were also blinded
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Experimental): Participants receive 8 mcg lubiprostone capsules twice daily (BID)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator): Participants receive 0 mcg capsules BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — 8 mcg administered orally twice daily (BID)
  Other Names: Amitiza
  Arms: Lubiprostone
Drug: Placebo — Matching placebo, 0 mcg administered orally twice daily (BID)
  Other Names: Matching Placebo
  Arms: Placebo

SUMMARY:
A study of the efficacy and safety of Lubiprostone in subjects diagnosed with IBS-M/IBS-U.

DETAILED DESCRIPTION:
To assess the efficacy and safety of oral lubiprostone, as compared to matching placebo, when administered orally (at 8 mcg twice daily [BID]) in subjects diagnosed with IBS-M/IBS-U.

ELIGIBILITY:
Inclusion Criteria:

* Subject meets the diagnosis of IBS-M or IBS-U as confirmed using the adapted ROME III Diagnostic Questionnaire for Adult Functional GI Disorders.
* Subject Screening diary entries must show an average worst abdominal pain in the past 24 hours score of at least 4 on a 11-point scale.
* Subject must be on a stable dose of selective serotonin re-uptake inhibitors (SSRIs), serotonin-specific reuptake inhibitor (SNRIs), or monoamine oxidase inhibitors (MAO) inhibitors if taking antidepressants.

Exclusion Criteria:

* Subject has current diagnosis of IBS with diarrhea (IBS-D) or IBS with constipation (IBS-C), according to Rome III Criteria.
* Any gastrointestinal (GI) condition, other than IBS-related, affecting GI motility or defecation.
* Medical/surgical condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, MD, Study Director — Mallinckrodt
Locations (16):
- United States (16):
  - E Squared Research, Inc., Huntsville, Alabama
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - GW Research Inc., Chula Vista, California
  - Inland Empire Liver Foundation, Rialto, California
  - Prestige Clinical Research Center, Miami, Florida
  - Advanced Gastroenterology Associates, LLC, Palm Harbor, Florida
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Charlotte, Concord, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Clinical Research Solutions, Jackson, Tennessee
  - Houston Endoscopy Research Center, Houston, Texas
  - Wellness Clinical Research Associates, McKinney, Texas
  - Advanced Clinical Research Associates, Plano, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants receive 0 mcg capsules twice daily (BID)
- Lubiprostone: Participants receive 8 mcg lubiprostone capsules BID
Period: Overall Study
Arm/Group | Placebo | Lubiprostone
Started | 34 | 37
Modified Intent to Treat (mITT) | 34 | 37
Safety Analysis Set (SAS) | 34 | 37
Completed | 33 | 30
Not Completed | 1 | 7
Not completed — Adverse Event | 0 | 4
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set (SAS), defined as all participants who take at least one dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Lubiprostone | Total
Number analyzed (Participants) | 34 | 37 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 34 | 65
  >=65 years | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 45 [21 to 71] | 49 [25 to 76] | 48 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 32 | 58
  Male | 8 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 26 | 33 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 37 | 71
Baseline Abdominal Pain [Mean (Standard Deviation); unit: units on a scale] — Participants rate their pain on a scale from 0-10, where 0=no pain and 10=the worst pain. A higher score means the pain is worse. Baseline is defined as the weekly average during the 4-week screening period.
  units on a scale | 5.90 (1.340) | 5.37 (1.406) | 5.62 (1.390)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Classified as an Overall Responder for Abdominal Pain
Description: An overall responder for abdominal pain is defined as a participant who is a weekly responder for at least 75% of observed treatment weeks.
Time Frame: within 12 weeks
Population: modified Intent to Treat (mITT), defined as all randomized subjects who take at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants | 10 | 11
Statistical Analysis 1: Comparison: Placebo vs Lubiprostone; P-value is from a Cochran-Mantel-Haenszel (CMH) test stratified by sex and baseline stool consistency; Test type: Other; p = 0.9870, Cochran-Mantel-Haenszel

2. Secondary Outcome: Number of Participants Classified as a Weekly Responder for Abdominal Pain
Description: Participants rate their pain on a pain intensity scale where 0=no pain and 10=worst pain. A higher score means the pain is worse.
  A weekly responder for abdominal pain is defined as a participant reporting ≥ 30% reduction from baseline in average of 24-hour worst abdominal pain scores for the preceding week.
Time Frame: within 12 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Week 1 | 7 | 7
  Week 2 | 13 | 8
  Week 3 | 11 | 12
  Week 4 | 13 | 19
  Week 5 | 15 | 18
  Week 6 | 16 | 15
  Week 7 | 14 | 14
  Week 8 | 11 | 18
  Week 9 | 13 | 15
  Week 10 | 15 | 12
  Week 11 | 14 | 14
  Week 12 | 10 | 12

3. Secondary Outcome: Number of Participants Classified as a Monthly Responder for Abdominal Pain
Description: A monthly responder for abdominal pain is defined as a participant who is a weekly responder for abdominal pain at least 2 of 4 weeks in the preceding month.
Time Frame: within 3 months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Month 1 | 12 | 14
  Month 2 | 16 | 16
  Month 3 | 15 | 13

4. Secondary Outcome: Number of Participants Classified as a Weekly Responder for Stool Consistency
Description: A weekly responder for stool consistency is defined as a participant having at least 50% reduction from baseline in percentage of days with extreme stool consistency for a given week.
Time Frame: within 12 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Week 1 | 5 | 12
  Week 2 | 6 | 11
  Week 3 | 5 | 10
  Week 4 | 7 | 10
  Week 5 | 11 | 9
  Week 6 | 8 | 7
  Week 7 | 8 | 9
  Week 8 | 6 | 9
  Week 9 | 6 | 5
  Week 10 | 8 | 10
  Week 11 | 7 | 6
  Week 12 | 8 | 8

5. Secondary Outcome: Number of Participants Classified as a Monthly Responder for Stool Consistency
Description: A monthly responder for stool consistency is defined as a participant who is a weekly responder for stool consistency at least 2 of 4 weeks in the preceding month.
Time Frame: within 3 months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Month 1 | 3 | 12
  Month 2 | 12 | 9
  Month 3 | 7 | 7

6. Secondary Outcome: Number of Participants Classified as an Overall Responder for Stool Consistency
Description: An overall responder for stool consistency is defined as a participant who qualifies as a weekly responder for stool consistency for at least 75% of observed treatment weeks.
Time Frame: within 3 months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants | 0 | 3

7. Secondary Outcome: Number of Participants Classified as a Weekly Responder for Irritable Bowel Syndrome (IBS) Symptoms
Description: A participant who achieves adequate relief of IBS symptoms during the preceding week is classified as a weekly responder for IBS symptoms.
Time Frame: within 12 weeks
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Week 1 | 14 | 9
  Week 2 | 16 | 14
  Week 3 | 18 | 15
  Week 4 | 21 | 20
  Week 5 | 22 | 19
  Week 6 | 19 | 17
  Week 7 | 16 | 17
  Week 8 | 17 | 20
  Week 9 | 18 | 14
  Week 10 | 15 | 15
  Week 11 | 18 | 14
  Week 12 | 4 | 6

8. Secondary Outcome: Number of Participants Classified as a Monthly Responder for IBS Symptoms
Description: A participant who is a weekly responder for IBS symptoms for at least 2 of the 4 weeks in the preceding month is classified as a monthly responder for IBS symptoms.
Time Frame: within 3 months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants
  Month 1 | 21 | 16
  Month 2 | 20 | 18
  Month 3 | 17 | 15

9. Secondary Outcome: Number of Participants Classified as an Overall Responder for IBS Symptoms
Description: A participant who is a weekly responder for IBS symptoms for at least 75% of observed treatment weeks is classified as an overall responder for IBS symptoms.
Time Frame: within 3 months
Population: mITT
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Lubiprostone
Number analyzed (Participants) | 34 | 37
Participants | 11 | 10

ADVERSE EVENTS:
Time Frame: 13 weeks
Description: Treatment-emergent adverse events, defined as any event with an onset date that is on or after the first dose of study medication and with an onset date no more than 7 days after the last dose of study medication.
Arm/Group | Placebo | Lubiprostone
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/34 | 1/37
Other Adverse Events (participants affected / at risk) | 8/34 | 12/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | Lubiprostone (N=37)
Colitis (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=34) | Lubiprostone (N=37)
Diabetic retinal oedema (Endocrine disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 4
Viral infection (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Mastitis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 0
Mean cell volume increased (Investigations) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes